CLINICAL TRIAL: NCT00704366
Title: A Phase I, Open-label, Dose-escalation Study to Assess the Safety and Tolerability of AZD0530 in Patients With Advanced Solid Malignancies
Brief Title: AZD0530 Study 21 - Phase I Study in Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Mary Stuart, BSc MSc MB BCh BAO MRCPI, Medical Science Director Emerging Oncology Product Team 1, AstraZeneca Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8180C00021
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Solid Tumor
Keywords: Advanced carcinoma
MeSH Terms: interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): AZD0530
  Interventions: Drug: AZD0530

INTERVENTIONS:
Drug: AZD0530 — oral, tablet, once daily, dose will be variable

SUMMARY:
This is a dose escalation study to assess the safety and tolerability of AZD0530 in patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced carcinoma / solid tumour of known primary site, which is refractory to standard therapies or for which no standard therapy exists
* World Health Organisation (WHO) performance status 0 to 2
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Inadequate bone marrow reserve
* Inadequate liver function, renal function or low hemoglobin
* Unresolved toxicity from anti-cancer therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the safety and tolerability of AZD0530 in Japanese patients with advanced solid malignancies by assessment of AEs, vital signs, ECG, laboratory findings, thoracic imaging and pulmonary function test. | Assessed on an ongoing basis after starting daily dosing with AZD0530

SECONDARY OUTCOMES:
To determine the single and multiple dose PK of AZD0530 when administered orally to patients with advanced solid malignancies by assessment of Cmin, Cmax, tmax, Cssmax, Cssmin, AUC0-t, AUC0-24, AUC, AUCss0-24, CL/F, t1/2 and R | 1 blood sample before the single dose and 11 samples afterwards until up to 146 hours after dose.1 blood sample before the start of daily dosing of AZD0530. With a further 12 samples over the next 22 days.
Tumor response | at entry and then 6 and 12 weeks after starting daily dosing of AZD0530. Assesments will then be made every 9 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Stuart, MD, Study Chair — AstraZeneca; Narikazu Boku, MD, Principal Investigator — Saint Marianna University School of Medicine
Locations (2):
- Japan (2):
  - Research Site, Takatsuk, Osaka
  - Research Site, Sunto-gun, Shizuoka

REFERENCES:
- [Derived] Fujisaka Y, Onozawa Y, Kurata T, Yasui H, Goto I, Yamazaki K, Machida N, Watanabe J, Shimada H, Shi X, Boku N. First report of the safety, tolerability, and pharmacokinetics of the Src kinase inhibitor saracatinib (AZD0530) in Japanese patients with advanced solid tumours. Invest New Drugs. 2013 Feb;31(1):108-14. doi: 10.1007/s10637-012-9809-7. Epub 2012 Mar 14. PMID 22415795